CLINICAL TRIAL: NCT03361410
Title: Examining the Impact of Grape Consumption on Brain Metabolism and Neuropsychological Performance in Patients Undergoing Neuroimaging Evaluation for Cognitive Decline: A Double-blinded Placebo Controlled Expansion Study
Brief Title: Impact of Grape Consumption on Brain Metabolism and Neuropsychological Performance Over 1 Year
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Daniel H. Silverman, Professor, Department of Molecular and Medical Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-001290
Record Dates: First submitted 2017-10-27; First posted 2017-12-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Decline in Cognition; Mild Cognitive Decline; Mild Cognitive Impairment; Dementia; Positron Emission Tomography (PET); F-18 Fluorodeoxyglucose (FDG); Cerebral Metabolism; Dietary Supplement; MCI; MDC; Grape; Memory; Randomized; Non-Drug; Supplement; Non-Pharmacologic; Natural; Red Wine; Free; UCLA; Brain Scan; Alzheimer's Disease; Brain Diseases; Central Nervous System Diseases; Cognition; Cognitive; Neurocognitive; Neurodegenerative
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Brain Diseases; Central Nervous System Diseases | interventions — whole grape extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grape Powder (Experimental)
  Interventions: Dietary Supplement: Grape Powder
- Placebo Powder (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Grape Powder — 36 g of grape powder to be taken twice/day (total of 72 g/day) for 12 months
  Arms: Grape Powder
Dietary Supplement: Placebo Powder — 36 g of placebo powder to be taken twice/day (total of 72 g/day) for 12 months
  Arms: Placebo Powder

SUMMARY:
Constituents of grapes have been studied for their antioxidant, anti-inflammatory, and anticarcinogenic properties. In the past decade, there has been emerging evidence regarding a potential role for grapes in slowing cognitive decline and other effects of aging. Furthermore, evidence has been obtained in vivo that supplementation with grape seed extract in aged rats improves cognitive performance, and that supplementation with grapes in people having decline in cognition leads to preservation of metabolism in brain regions important to cognitive function over a period of six months. The investigator aims to measure effects of grape intake on cerebral metabolism and neuropsychological performance, and to determine whether initial patterns, and magnitude of change, of cerebral metabolism assessed by positron emission tomography (PET) can serve respectively as a predictor of, and biomarker for, the magnitude of cognitive changes resulting from intake of grapes over a period of at least one year.

DETAILED DESCRIPTION:
As the number of people age 65 years old or older continues to increase, population aging has a profound impact on healthcare systems, and specifically the emergence of dementia in literally epidemic proportions. Numerous studies on the associations between grape consumption and dementia and Alzheimer's disease have found evidence to support the use of grapes and grape products as a safe and effective way to treat and delay the onset of dementia. For the present study, the Investigator aims (1) to identify regional cerebral metabolic changes associated with grape intake, (2) to determine whether the presence and magnitude of therapeutic responses to grape in patients undergoing neuroimaging evaluation for cognitive decline can be predicted by particular patterns of regional brain metabolism, and (3) to statistically assess the relationships between brain metabolism assessed by PET and cognitive function in randomized experimental arms. A total of 32 patients from a community sample of patients referred to UCLA NeuroPET Clinics by their neurologists for further evaluation by brain imaging will be studied in this placebo-controlled, double-blinded study. Subjects who have met the screening criteria will be randomized to receive 72 g of grape powder or placebo, reconstituted in water, per day. Regional brain metabolism will be measured with a PET scanner, and cognitive function will be measured by a neuropsychologic test battery assessed at baseline, 6 months following initiation of consumption, and 1 year following initiation of consumption of the grapes of placebo formulation.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the UCLA NeuroPET Clinics for concern of cognitive decline and/or behavioral changes.
* Standard history, physical, and laboratory screen performed to identify possible presence of depression, substance abuse, malnourishment, medical effects and interactions, cardiopulmonary compromise, electrolyte/calcium imbalance, anemia, hypoxemia, infection, thyroid dysfunction, renal dysfunction, hepatic dysfunction, or glucose dysregulation, and appropriate therapies administered (if any).
* Appropriate neurological consultation has been obtained, as well as CT/MRI and/or neurosurgical consultation if history or neurologic exam reveal findings suspicious for stroke, tumor, bleed, ictal activity, or hydrocephalus.

Exclusion Criteria:

* Subjects under age 65 and over age 85, in order to enhance the clinical relevance of the project by focusing on the age groups in whom serious concerns about early signs and symptoms of senile onset dementia are most typically emerging.
* Have begun cholinesterase inhibitors or memantine in the last 6 months.
* Patient lacks adequate functional status and/or caregiver support to reliably follow grape consumption regimen.
* Claustrophobia or other condition that would preclude PET from being acquired, or visual, auditory, language, or motor deficits that would preclude accurate neuropsychological testing.
* Non-English speaking subjects, due to lack of neuropsychologic testing or equivalent instruments in non-English languages.
* Subjects with a history of allergy to grapes or grape products.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Regional Cerebral Metabolism | Baseline and 12 months
  Changes from baseline in regional cerebral metabolism

SECONDARY OUTCOMES:
Changes in neuropsychological performance measures | Baseline, 6 months, and 12 months
  Changes in cognitive performance over time within each group will be measured through the neuropsychological assessments listed below, as administered by trained psychometrists under direct supervision of a licensed neuropsychologist, and will be correlated with changes in regional cerebral metabolism.
Changes in neuropsychological performance measures: Mini-Mental State Examination | Baseline, 6 months, and 12 months
  Mini-Mental State Examination (Folstein, 1975)
Changes in neuropsychological performance measures: Wechsler Adult Intelligence Scale (WAIS-III) Digit Span | Baseline, 6 months, and 12 months
  Wechsler Adult Intelligence Scale (WAIS-III) Digit Span (Wechsler, 1997)
Changes in neuropsychological performance measures: Trail Making Test Part B | Baseline, 6 months, and 12 months
  Trail Making Test Part B (Reitan, 1958)
Changes in neuropsychological performance measures: Functional Activities Questionnaire | Baseline, 6 months, and 12 months
  Functional Activities Questionnaire (Pfeffer et al., 1982)
Changes in neuropsychological performance measures: Verbal Memory | Baseline, 6 months, and 12 months
  NeuroTrax BrainCare, a cloud-based computer application that includes a series of tests and associated reports, will be used to measure Verbal Memory.
Changes in neuropsychological performance measures: Non-Verbal Memory | Baseline, 6 months, and 12 months
  Non-Verbal Memory (measured using the NeuroTrax BrainCare application)
Changes in neuropsychological performance measures: Verbal Function | Baseline, 6 months, and 12 months
  Verbal Function (measured using the NeuroTrax BrainCare application)
Changes in neuropsychological performance measures: Stroop Interference | Baseline, 6 months, and 12 months
  Stroop Interference (measured using the NeuroTrax BrainCare application)
Changes in neuropsychological performance measures: Problem Solving | Baseline, 6 months, and 12 months
  Problem Solving (measured using the NeuroTrax BrainCare application)
Changes in neuropsychological performance measures: Visual Spatial Processing | Baseline, 6 months, and 12 months
  Visual Spatial Processing (measured using the NeuroTrax BrainCare application)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Silverman, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States